CLINICAL TRIAL: NCT04320069
Title: Evaluating the Safety and Effectiveness of the Omnipod Horizon™ CGM-informed Bolus Calculator in Patients With Type 1 Diabetes
Brief Title: Continuous Glucose Monitoring System (CGM)-Informed Bolus Calculator Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G200018
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Type 1 Diabetes
Keywords: T1D; Omnipod
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This is a single-arm, multi-center, prospective clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Omnipod Horizon™ Automated Glucose Control System (Experimental): All subjects using the Omnipod Horizon™ Automated Glucose Control System in Manual Mode without a connected CGM for 7 days and with a connected CGM for 7 days.
  Interventions: Device: Omnipod Horizon™ Automated Glucose Control System

INTERVENTIONS:
Device: Omnipod Horizon™ Automated Glucose Control System — Omnipod Horizon™ Automated Glucose Control System use in Manual Mode

SUMMARY:
Subjects will use the Omnipod Horizon™ System in Manual Mode in an outpatient setting for 14-days. Subjects will be trained to use the Manual Mode feature of the Omnipod Horizon™ System including how to use the bolus calculator using manual entry of blood glucose values or by using the CGM-informed bolus calculator.

DETAILED DESCRIPTION:
The study schedule consists of two outpatient phases:

1. 7 days of Omnipod Horizon™ use in Manual Mode without a connected CGM using manual entry of BG values to deliver boluses (Phase 1) followed by;
2. 7 days of Omnipod Horizon™ use in Manual Mode with a connected CGM using the CGM-informed bolus calculator to deliver boluses (Phase 2)

Following subject screening, system training and enrollment, subjects will commence the first 7-day Manual Mode phase of the study.

Subjects will be trained to use the Manual Mode feature of the system including how to use the bolus calculator using manual entry of BG values or by using the CGM-informed bolus calculator.

After completion of the first 7 days of the Manual Mode phase using the Omnipod Horizon™ without a connected CGM, subjects will transition to the next 7 days of the Manual Mode phase using the system with a connected CGM using the CGM-informed bolus calculator to deliver boluses.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent/assent 2-70 years
2. Subjects aged < 18 years must be living with parent/legal guardian
3. Diagnosed with type 1 diabetes for at least 6 months. Diagnosis is based on investigator's clinical judgment
4. Must be a current Omnipod user, or have used an Omnipod in the past
5. Investigator has confidence that the subject, parent, or legal guardian, can successfully operate all study devices and can adhere to the protocol
6. Willing to use only the following types of Insulin during the study: Humalog, Novolog, Admelog, or Apidra
7. Must be willing to use the Omnipod Horizon™ in Manual Mode only and agree not to use Automated Mode functionality
8. Must be willing to use the Omnipod Horizon™ bolus calculator without a connected CGM for the first 7-days of Manual Mode (Phase 1) while manually entering BG values to deliver boluses
9. Must be willing to use the Omnipod Horizon™ bolus calculator with a connected CGM for the last 7-days of Manual Mode (Phase 2) using the CGM-informed bolus calculator to deliver boluses
10. Willing to wear the system continuously throughout the study
11. For subjects not currently enrolled in the Omnipod Horizon™ Pivotal Study (G190270), A1C <10%
12. Must be willing to use the Dexcom App on the Omnipod Horizon™ PDM as the sole source of Dexcom data (except for the Dexcom Follow App)
13. Able to read and speak English fluently (if subject is a young child then Caregiver must meet the criteria)
14. Willing and able to sign the Informed Consent Form (ICF) and/or has a parent/guardian willing and able to sign the ICF. Assent will be obtained from subjects aged < 18 years per State requirements.
15. For subjects aged 2-5.9 years of age, parents or trained caregivers agree to be physically present during the decision and delivery of insulin boluses for this age group, as well as agree to be available for glucose monitoring and treatment during the 4-hour post bolus period.

Exclusion Criteria:

1. A medical condition, which in the opinion of the investigator, would put the subject at an unacceptable safety risk
2. History of severe hypoglycemia in the past 6 months
3. History of DKA in the past 6 months, unrelated to an intercurrent illness or infusion set failure
4. Plans to receive blood transfusion over the course of the study
5. Currently diagnosed with anorexia nervosa or bulimia
6. Acute or chronic kidney disease or currently on hemodialysis
7. History of adrenal insufficiency
8. Has taken oral or injectable steroids within the past 8 weeks or plans to take oral or injectable steroids during the study
9. Unable to tolerate adhesive tape or has any unresolved skin condition in the area of sensor or pump placement
10. Plans to use insulin other than U-100 insulin intended for use in the study device during the study
11. Use of non-insulin anti-diabetic medication other than metformin (e.g. GLP1 agonist, SGLT2 inhibitor, DPP-4 inhibitor, pramlintide)
12. Current or known history of coronary artery disease that is not stable with medical management, including unstable angina, or angina that prevents moderate exercise despite medical management, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the previous 12 months
13. Clinical signs of hypothyroidism and hyperthyroidism
14. Pregnant or lactating, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD or implant)
15. Currently participating or plans to participate in another clinical study using an investigational drug or device other than Omnipod Horizon™. Subjects may be recruited from the Omnipod Horizon Pivotal Study (G190270) prior to their recommencement of the pivotal study after study pause.
16. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the investigator's clinical judgment

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Pinsker, MD, Study Chair — Sansum Diabetes Research Institute
Locations (4):
- United States (4):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - University of Colorado Denver, Denver, Colorado
  - Atlanta Diabetes, Atlanta, Georgia
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinsker JE, Church MM, Brown SA, Voelmle MK, Bode BW, Narron B, Huyett LM, Lee JB, O'Connor J, Benjamin E, Dumais B, Ly TT. Clinical Evaluation of a Novel CGM-Informed Bolus Calculator with Automatic Glucose Trend Adjustment. Diabetes Technol Ther. 2022 Jan;24(1):18-25. doi: 10.1089/dia.2021.0140. Epub 2021 Sep 3. PMID 34491825

RESULTS

PARTICIPANT FLOW:
Period: Phase 1: Omnipod Horizon™ Without CGM
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Started | 25
Completed | 25
Not Completed | 0
Period: Phase 2: Omnipod Horizon™ With CGM
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.8 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time <70 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1 (comparing the 4-hour post bolus period)
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Phase 1 | 2.8 (2.7)
  Phase 2 | 2.1 (2.0)

2. Primary Outcome: Percentage of Time >180 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1 (comparing the 4-hour post bolus period)
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Phase 1 | 32.1 (15.7)
  Phase 2 | 34.0 (16.0)

3. Secondary Outcome: Mean Glucose
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1 (comparing the 4-hour post bolus period)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
mg/dL
  Phase 1 | 158.7 (21.3)
  Phase 2 | 163.3 (23.6)

4. Secondary Outcome: Percentage of Time <54 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1 (comparing the 4-hour post bolus period)
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Phase 1 | 0.5 (1.0)
  Phase 2 | 0.3 (0.7)

5. Secondary Outcome: Percentage of Time ≥ 250 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1 (comparing the 4-hour post bolus period)
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Phase 1 | 8.2 (6.9)
  Phase 2 | 9.7 (10.3)

6. Secondary Outcome: Percentage of Time ≥ 300 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1 (comparing the 4-hour post bolus period)
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Phase 1 | 2.0 (2.6)
  Phase 2 | 2.6 (3.7)

7. Secondary Outcome: Percentage of Time in Range 70-180 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1 (comparing the 4-hour post bolus period)
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Phase 1 | 65.1 (15.4)
  Phase 2 | 63.8 (15.7)

8. Secondary Outcome: Mean Glucose
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1, during the day (6AM up to 12AM), overnight (12AM up to 6AM), and overall
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
mg/dL
  Day Time Phase 1 | 150.1 (18.1)
  Day Time Phase 2 | 152.8 (20.7)
  Night Time Phase 1 | 151.4 (27.7)
  Night Time Phase 2 | 155.6 (28.3)
  Overall Phase 1 | 150.4 (18.9)
  Overall Phase 2 | 153.5 (20.3)

9. Secondary Outcome: Percentage of Time <54 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1, during the day (6AM up to 12AM), overnight (12AM up to 6AM), and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Day Time Phase 1 | 0.5 (0.8)
  Day Time Phase 2 | 0.3 (0.7)
  Night Time Phase 1 | 0.3 (0.9)
  Night Time Phase 2 | 0.4 (0.7)
  Overall Phase 1 | 0.4 (0.7)
  Overall Phase 2 | 0.4 (0.5)

10. Secondary Outcome: Percentage of Time <70 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1, during the day (6AM up to 12AM), overnight (12AM up to 6AM), and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Day Time Phase 1 | 2.9 (2.7)
  Day Time Phase 2 | 2.7 (2.2)
  Night Time Phase 1 | 2.8 (4.1)
  Night Time Phase 2 | 2.7 (3.7)
  Overall Phase 1 | 2.9 (2.3)
  Overall Phase 2 | 2.7 (2.0)

11. Secondary Outcome: Percentage of Time >180 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1, during the day (6AM up to 12AM), overnight (12AM up to 6AM), and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Day Time Phase 1 | 25.9 (13.5)
  Day Time Phase 2 | 26.8 (14.2)
  Night Time Phase 1 | 26.9 (18.9)
  Night Time Phase 2 | 26.9 (19.0)
  Overall Phase 1 | 26.2 (13.7)
  Overall Phase 2 | 26.8 (14.0)

12. Secondary Outcome: Percentage of Time ≥ 250 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1, during the day (6AM up to 12AM), overnight (12AM up to 6AM), and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Day Time Phase 1 | 6.3 (4.9)
  Day Time Phase 2 | 7.0 (8.3)
  Night Time Phase 1 | 6.3 (8.3)
  Night Time Phase 2 | 8.2 (11.2)
  Overall Phase 1 | 6.3 (5.1)
  Overall Phase 2 | 7.3 (7.4)

13. Secondary Outcome: Percentage of Time ≥ 300 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1, during the day (6AM up to 12AM), overnight (12AM up to 6AM), and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Day Time Phase 1 | 1.4 (1.9)
  Day Time Phase 2 | 1.9 (2.8)
  Night Time Phase 1 | 1.5 (3.4)
  Night Time Phase 2 | 1.8 (3.5)
  Overall Phase 1 | 1.4 (1.8)
  Overall Phase 2 | 1.8 (2.3)

14. Secondary Outcome: Percentage of Time in Range 70-180 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1, during the day (6AM up to 12AM), overnight (12AM up to 6AM), and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Day Time Phase 1 | 71.1 (13.4)
  Day Time Phase 2 | 70.6 (14.3)
  Night Time Phase 1 | 70.3 (17.2)
  Night Time Phase 2 | 70.4 (18.8)
  Overall Phase 1 | 70.9 (13.2)
  Overall Phase 2 | 70.6 (14.1)

15. Secondary Outcome: Percentage of Time in Range 70-140 mg/dL
Description: Glucose metric from continuous glucose monitoring system (CGM)
Time Frame: Phase 2 compared to Phase 1, during the day (6AM up to 12AM), overnight (12AM up to 6AM), and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent Time in Range
  Day Time Phase 1 | 47.4 (13.9)
  Day Time Phase 2 | 45.8 (15.2)
  Night Time Phase 1 | 46.5 (18.1)
  Night Time Phase 2 | 42.1 (18.5)
  Overall Phase 1 | 47.2 (13.8)
  Overall Phase 2 | 44.9 (14.8)

16. Secondary Outcome: Standard Deviation
Description: Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the standard deviation (SD)
Time Frame: Phase 2 compared to Phase 1, during the day (6AM up to 12AM), overnight (12AM up to 6AM), and overall
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
mg/dL
  Day Time Phase 1 | 52.1 (12.2)
  Day Time Phase 2 | 51.4 (12.8)
  Night Time Phase 1 | 47.3 (15.6)
  Night Time Phase 2 | 47.2 (16.7)
  Overall Phase 1 | 51.9 (12.1)
  Overall Phase 2 | 51.6 (12.8)

17. Secondary Outcome: Coefficient of Variation
Description: Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the coefficient of variation (CV)
Time Frame: Phase 2 compared to Phase 1, during the day (6AM up to 12AM), overnight (12AM up to 6AM), and overall
Measure: Mean (Standard Deviation); unit: Percent coefficient of variation
Arm/Group | Omnipod Horizon™ Automated Glucose Control System
Number analyzed (Participants) | 25
Percent coefficient of variation
  Day Time Phase 1 | 34.6 (6.6)
  Day Time Phase 2 | 33.5 (6.7)
  Night Time Phase 1 | 31.0 (7.1)
  Night Time Phase 2 | 30.0 (8.0)
  Overall Phase 1 | 34.3 (5.8)
  Overall Phase 2 | 33.4 (6.3)

ADVERSE EVENTS:
Time Frame: First day of Phase 1 to last day of Phase 2, an average of 14 days.
Groups:
- Single: All subjects using the Omnipod Horizon™ Automated Glucose Control System in Manual Mode without a connected CGM for 7 days and with a connected CGM for 7 days.
  Omnipod Horizon™ Automated Glucose Control System: Omnipod Horizon™ Automated Glucose Control System use in Manual Mode
Arm/Group | Single
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single (N=25)
Pyelonephritis (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT04320069/Prot_SAP_001.pdf